CLINICAL TRIAL: NCT04876625
Title: Effects of myTAP Oral Appliance Therapy on Cardio-respiratory Dynamics in Mouth-breathers Who Snore
Brief Title: OA Therapy for Mouth-breathers Who Snore
Acronym: OATMB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Emet D. Schneiderman, PhD, Professor, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB2019-0421
Record Dates: First submitted 2021-04-29; First posted 2021-05-06 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Snoring; Mouth Breathing; Obstructive Sleep Apnea
Keywords: oral appliance; mouth shield; snoring
MeSH Terms: conditions — Snoring; Mouth Breathing; Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Single center, randomized trial using a parallel group design
Who Masked: Outcomes Assessor
Masking Description: Investigators scoring sleep studies and doing data analysis will be blinded with regard to group identity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- OA plus MS 8wk (Experimental): Oral Appliance plus Mouth Shield for 8-weeks
  Interventions: Device: myTAP oral appliance plus mouth shield
- OA Alone 4wk (Active Comparator): Oral Appliance is used alone for first 4 weeks followed by 4 weeks of Oral Appliance plus Mouth Shield
  Interventions: Device: myTAP oral appliance alone for first 4 weeks

INTERVENTIONS:
Device: myTAP oral appliance plus mouth shield — myTAP anti-snoring oral appliance worn with mouth shield for all 8-weeks; the mouth shield is a comfort accessory that fits over the oral appliance itself and extends into the oral vestibule.
  Other Names: anti-snoring device; midline traction oral appliance
  Arms: OA plus MS 8wk
Device: myTAP oral appliance alone for first 4 weeks — myTAP anti-snoring oral appliance worn alone for first 4 weeks followed by wearing it for 4 weeks with the mouth shield
  Other Names: anti-snoring device; midline traction oral appliance
  Arms: OA Alone 4wk

SUMMARY:
Breathing is one of the body's vital functions that occur under normal conditions using the nose. When humans breathe primarily through the mouth instead of the nose, this is referred to as mouth breathing. Snoring and obstructive sleep apnea (OSA) occur frequently in mouth breathers. Mouth breathing impairs oral health, reduces quantity and quality of saliva, and increases dry mouth, risk of developing dental caries, gingival inflammation, bad breath and dry lips. Serious health conditions associated with an obstructed upper airway in those who snore include hypertension, cardiovascular disease and mild cognitive impairment.

Oral appliances (OAs) that bring the lower jaw (mandible) forward have been shown to be highly effective in reducing snoring and interruptions in breathing (respiratory events) that occur in those who snore and/or have OSA. The myTAP™ OA (AMI, Dallas, TX) includes an optional mouth shield (MS) that is anticipated to promote nasal breathing. The purpose of this study is to investigate the effects of oral appliance plus mouth shield therapy on sleep cardio-respiratory dynamics (breathing and heart activity) and their effect on improving OSA and oral health, especially of the periodontal tissues, in confirmed mouth breathers who snore and/or have OSA. As many as 70 adults at least 18 years old will be recruited to participate.

All participants will wear the OA during sleep for 8 weeks (Phase 1). Half of the participants will be randomly assigned to wear the OA only for the first 4 weeks; all will wear both the OA and MS for the last 4 weeks. Participants will wear an easy-to-use home sleep recording system (NOX T3) for 2 nights at the start of the study and again at 4 weeks and 8 weeks. Based on the investigators' experience, some participants will not have achieved maximal benefit from the OA at 8 weeks, and will require addition adjustment. These participants will enter a second phase of the study where they will have 1 or more sleep studies done at 2 week intervals, and will further adjust their OAs (that is, advance the mandible) to eliminate snoring.

DETAILED DESCRIPTION:
Background: Respiration is one of the body's vital functions that occurs under normal conditions using the nose. When nasal breathing is supplemented by or supplanted through the mouth, this is referred to as mouth breathing. Primary snoring and obstructive sleep apnea (OSA) are frequent findings in mouth breathers, regardless of age. In children, mouth breathing is often associated with enlarged adenoids and tonsils, changes in body posture, hyperactivity, attention deficit and impaired learning. In all ages, mouth breathing impairs oral health, reduces quantity and quality of saliva, and increases dry mouth, risk of developing dental caries, gingival inflammation, bad breath and dry lips. Symptoms associated with an obstructed upper airway in those who snore include hypertension, cardiovascular disease and mild cognitive impairment. There are currently no data on the effects of oral appliance plus mouth shield therapy on sleep cardio-respiratory dynamics and their effect on improving OSA and oral health, especially periodontal health, in mouth breathers.

Methods: Evaluation of the effects of the FDA cleared MyTAP midline traction type oral appliance (OA; AMI, Dallas, TX) in combination with its FDA-cleared mouth shield (MS) in treating confirmed mouth breathers who snore and/or have OSA.

Power analysis: Sample size (n=40) is based on a-posteriori power of 80% observed in the investigative team's recently completed randomized controlled trial (RCT) comparing two OA designs. As many as 70 participants will be enrolled to account for drop-outs.

Design: Single center, prospective randomized clinical trial using a parallel group design.

Randomization: Using an online randomizer software, half of the subjects will be assigned to Group "OA plus MS 8wk", OA use with MS for 8-weeks and group "OA Alone 4wk" (no MS) for first 4-weeks. The OA Alone 4wk group will add MS use after 4-weeks and continue to use the combination for subsequent 4-weeks.

Clinically standard periodontal exams will be performed at baseline (T0), after 4-weeks (T2) and after 8 weeks (T3). The dentist-fitted OA will be applied chair-side and adjusted to a starting position of 60% of the lower jaw's maximum comfortable protrusion. All participants will wear the OA nightly during sleep for 8-consecutive weeks. Subjects will be instructed to advance the jaw up to 0.5 mm every 2 nights (less frequently if needed to minimize transient discomfort). Subjects will use the EverSleep Wearable Sleep Tracker app (Somno Health Inc., Golden CO) on their smart phones to monitor their own snoring nightly, and self-titrate their OAs until no snore detection is reported by the software.

Based on the investigators' recently completed study (IRB2017-0390) and another study published on this kind of appliance, some participants will not have achieved maximal benefit from the OA, and will require addition adjustment. These participants will enter Phase 2 of the study where they will have 1 or 2 more sleep studies done at 2 week intervals, and will further adjust their OAs (that is, advance their lower jaws) to eliminate snoring.

The investigators will evaluate differences in sleep respiration events, snoring and other measures at all time points except T1. Periodontal exams (gums and supporting tissues) will be performed at T1-T3 and T5. Comparison will be done between and within group (that is, with and without the MS) .

The purpose of collecting sleep data with OA use is to determine its success in promoting stable respiration during sleep and reducing the number of events in which breathing stops (apneas) or diminished (hypopneas) and the amount of oxygen in the blood is low (oxygen desaturation).

The sleep recorder (NOX T3, Nox Medical , Reykjavík, Iceland) is a Food and Drug Administration (FDA) cleared and certified for sale within the European Economic area (CE marked). The midline traction oral appliance (myTAP, AMI Inc., Dallas Texas) is currently marketed as a medical device to treat snoring and obstructive sleep apnea and is FDA cleared and CE marked. The EverSleep device (Somnohealth, Golden Colorado) is a wearable sleep coaching device and is not an FDA 510(k) cleared medical device.

ELIGIBILITY:
Inclusion Criteria

1. At least 18 years old (adults & seniors, male & female).
2. Presence of snoring, mouth-breathing or previously diagnosed with obstructive sleep apnea.
3. If present, stable cardiopulmonary disease (heart failure, chronic obstructive pulmonary disease, ventricular dysrhythmia), morbid obesity or other serious health conditions, must be under a physician's care; participant must obtain written permission from the physician to participate in this study.
4. If participated in recent OA clinical trial at the Texas A&M University College of Dentistry (IRB# 2017-0390) must be willing to try the myTAP as alternative to OA that is currently being used. The myTAP is a chairside-fitted OA that may be more comfortable and effective than the previous OAs and includes a mouth-shield.
5. At least 8 teeth per arch to support OA device.
6. Mallampati score from I to III; palatine tonsils grade 0,1 or 2.
7. Willing & able to provide verbal & written informed consent in English & understand how to apply, remove & utilize the sleep recorder & the OA device, as well as fill out brief questionnaires & nightly sleep diary.

Exclusion Criteria:

1. Unable or unwilling to complete the study demands & schedule.
2. Active temporomandibular joint dysfunction (TMD) or jaw muscle pain, morphological airway abnormalities.
3. Severe restrictions in jaw opening.
4. Pre-existing difficulty swallowing; throat or neck related health issues; unmanaged endocrine dysfunction.
5. Severe chronic nasal obstruction that precludes possibility of nasal breathing.
6. Severe psychiatric & neurological disorders; intellectually disabled.
7. Advanced periodontal disease (e.g., loose teeth).
8. History of uvulopalatopharyngoplasty (UPPP) surgery.
9. Loose teeth, loose crowns or fillings.
10. Removable dentures or bridges.
11. Temporary crowns.
12. Orthodontic braces.
13. Other oral conditions which would be adversely affected by wearing dental appliances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2021-09-25 (Actual); Study Completion 2022-09-25 (Actual)

PRIMARY OUTCOMES:
Respiratory Event Index (REI) at T2 | 4 weeks
  Number of apneas and hypopneas per hour of recording using the NOX T3 sleep recording system at T2 (4 weeks).
  REI is reported instead of Apnea Hypopnea Index (AHI), as it is a more appropriate measure for home sleep testing. Apneas are scored when there is a 90% drop in the flow signal between 10 and 120 seconds. Hypopneas are scored when there is a 30% drop in flow signal between 10 and 120 seconds followed by either a drop in oxygen saturation or an arousal.

CONTACTS AND LOCATIONS:
Overall Officials: Emet Schneiderman, PhD, Principal Investigator — Texas A&M University College of Dentistry
Locations (1):
- Texas A&M University College of Dentistry, Dallas, Texas, United States

REFERENCES:
- [Background] Hoekema A, Doff MH, de Bont LG, van der Hoeven JH, Wijkstra PJ, Pasma HR, Stegenga B. Predictors of obstructive sleep apnea-hypopnea treatment outcome. J Dent Res. 2007 Dec;86(12):1181-6. doi: 10.1177/154405910708601208. PMID 18037652

DOCUMENTS (1):
  • Informed Consent Form (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/25/NCT04876625/ICF_000.pdf